CLINICAL TRIAL: NCT03697486
Title: The Effect of Breakfast With Different Macronutrient Composition on PYY, Ghrelin, GLP-1, Glucose Level, VAS for Hunger, VAS for Satiety and Ad Libitum Intake 4 Hours After Breakfast in Obese Women
Brief Title: The Effect of Breakfast With Different Macronutrient Composition on PYY, Ghrelin, GLP-1,Glucose Level, VAS for Hunger, VAS for Satiety and Ad Libitum Intake 4 Hours After Breakfast in Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: SEAMEO Regional Centre for Food and Nutrition (Other); Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Fiastuti Witjaksono, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GuthormonesS3
Record Dates: First submitted 2018-10-02; First posted 2018-10-05 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: PYY; Ghrelin; Appetite; Gut Hormones; Obesity; Protein Consumption
Keywords: PYY; ghrelin; ad libitum intake; high protein diet; moderately protein diet; low protein diet; breakfast; obesity
MeSH Terms: conditions — Obesity | interventions — Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Protein (Experimental): (40,6% protein)
  Interventions: Behavioral: diet with different composition
- Moderate Protein (Experimental): (23.5% protein)
  Interventions: Behavioral: diet with different composition
- Low Protein (Experimental): (12.4% protein)
  Interventions: Behavioral: diet with different composition

INTERVENTIONS:
Behavioral: diet with different composition — Participants should not eat within the last 10 hours. Participants could drink mineral water up to 2 hours before intervention. Breakfast given is a milk-based formula which has to be finished within 15 minutes, and subjects could only consume 600 mL of mineral water within the next 4 hours after intervention. Participants' blood was taken before intervention, and 15, 60, 120, and 180 minutes after intervention, then examined in laboratory to measure ghrelin and PYY level. Breakfast given is adjusted to participants' energy requirement. Energy requirement is calculated by adding basal metabolic rate (BMR) with additional energy from physical activity. Different composition of protein, carbohydrate and fat were given to each arm depends on their group.
  After 4 hours, participants were given ad libitum meal. After the participants done eating, the calorie in meal taken by participants was measured.

SUMMARY:
Gut hormones, such as PYY and ghrelin, are associated with appetite control and obesity. Protein is thought to be the most satieting nutrient and could affect production of several gut hormones. This study's objective is to find the effect of breakfast with different protein composition on PYY, ghrelin, and ad libitum intake four hours after breakfast.

The research methodology was used a clinical trial with 22 obese women participants. Subjects were given three types of breakfast: low protein consumption (12.4% protein), medium protein (23.5% protein), and high protein (40,6% protein). PYY and ghrelin level were measured at 0, 15, 60, 120, and 180 minutes after breakfast. Ad libitum meal was given four hours after breakfast and measured after.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-30 (obese)
* with stable body weight within the last 6 months (body weight change less than 4 kg)
* normal blood glucose level.

Exclusion Criteria:

* patients who never had breakfast
* patients in weight loss program
* patients consuming lipid-absorption inhibitor or appetite-suppressing drugs
* patients that have had gastrointestinal tract resection.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Ghrelin levels at 0 minute | baseline
  analyzed by ELISA, directly taken after having the breakfast with different protein composition
Ghrelin levels at 15 minute | 15 minutes
  analyzed by ELISA, taken 15 minutes after having the breakfast with different protein composition
Ghrelin levels at 60 minute | 60 minutes
  analyzed by ELISA, taken 60 minutes after having the breakfast with different protein composition
Ghrelin levels at 120 minute | 120 minutes
  analyzed by ELISA, taken 60 minutes after having the breakfast with different protein composition
Ghrelin levels at 180 minute | 180 minutes
  analyzed by ELISA, taken 60 minutes after having the breakfast with different protein composition
PYY levels at 0 minute | baseline
  analyzed by Radioimmunoassay, directly taken after having the breakfast with different protein composition
PYY levels at 15 minute | 15 minutes
  analyzed by Radioimmunoassay, taken 15 minutes after having the breakfast with different protein composition
PYY levels at 60 minute | 60 minutes
  analyzed by Radioimmunoassay, taken 60 minutes after having the breakfast with different protein composition
PYY levels at 120 minute | 120 minutes
  analyzed by Radioimmunoassay, taken 120 minutes after having the breakfast with different protein composition
PYY levels at 180 minute | 180 minutes
  analyzed by Radioimmunoassay, taken 180 minutes after having the breakfast with different protein composition
GLP-1 levels at 0 minute | baseline
  analyzed by ELISA, directly taken after having the breakfast with different protein composition
GLP-1 levels at 15 minute | 15 minutes
  analyzed by ELISA, taken 15 minutes after having the breakfast with different protein composition
GLP-1 levels at 60 minute | 60 minutes
  analyzed by ELISA, taken 60 minutes after having the breakfast with different protein composition
GLP-1 levels at 120 minute | 120 minutes
  analyzed by ELISA, taken 120 minutes after having the breakfast with different protein composition
GLP-1 levels at 180 minute | 180 minutes
  analyzed by ELISA, taken 180 minutes after having the breakfast with different protein composition
Glucose levels at 0 minute | baseline
  analyzed by standard random glucose level from venous blood, taken directly after having the breakfast with different protein composition
Glucose levels at 15 minute | 15 minutes
  analyzed by standard random glucose level from venous blood, taken 15 minutes after having the breakfast with different protein composition
Glucose levels at 60 minute | 60 minutes
  analyzed by standard random glucose level from venous blood, taken 60 minutes after having the breakfast with different protein composition
Glucose levels at 120 minute | 120 minutes
  analyzed by standard random glucose level from venous blood, taken 120 minutes after having the breakfast with different protein composition
Glucose levels at 180 minute | 180 minutes
  analyzed by standard random glucose level from venous blood, taken 180 minutes after having the breakfast with different protein composition
Ad Libitum intake | 4 hours
  Mean Ad Libitum intake (calories) in subjects four hours after breakfast with different protein composition
VAS for hunger at 0 minutes | baseline
  Visual Analog Scale, a scale in the form of an empty straight line with no values but only several level point (ex: if the line is 10cm, then each cm represent 1 level). Extreme choices are both ends of the straight line. The minimum value is at the left end and the maximum value is at the right end. The subject must make a choice between the two ends of the line by giving an X mark (ex : if the subject feels less hunger, then the subject should mark X at the second point from far left), directly taken after having the breakfast with different protein composition
VAS for hunger at 15 minutes | 15 minutes
  Visual Analog Scale, a scale in the form of an empty straight line with no values but only several level point (ex: if the line is 10cm, then each cm represent 1 level). Extreme choices are both ends of the straight line. The minimum value is at the left end and the maximum value is at the right end. The subject must make a choice between the two ends of the line by giving an X mark (ex : if the subject feels less hunger, then the subject should mark X at the second point from far left), taken 15 minutes after having the breakfast with different protein composition
VAS for hunger at 60 minutes | 60 minutes
  Visual Analog Scale, a scale in the form of an empty straight line with no values but only several level point (ex: if the line is 10cm, then each cm represent 1 level). Extreme choices are both ends of the straight line. The minimum value is at the left end and the maximum value is at the right end. The subject must make a choice between the two ends of the line by giving an X mark (ex : if the subject feels less hunger, then the subject should mark X at the second point from far left), taken 60 minutes after having the breakfast with different protein composition
VAS for hunger at 120 minutes | 120 minutes
  Visual Analog Scale, a scale in the form of an empty straight line with no values but only several level point (ex: if the line is 10cm, then each cm represent 1 level). Extreme choices are both ends of the straight line. The minimum value is at the left end and the maximum value is at the right end. The subject must make a choice between the two ends of the line by giving an X mark (ex : if the subject feels less hunger, then the subject should mark X at the second point from far left), taken 120 minutes after having the breakfast with different protein composition
VAS for hunger at 180 minutes | 180 minutes
  Visual Analog Scale, a scale in the form of an empty straight line with no values but only several level point (ex: if the line is 10cm, then each cm represent 1 level). Extreme choices are both ends of the straight line. The minimum value is at the left end and the maximum value is at the right end. The subject must make a choice between the two ends of the line by giving an X mark (ex : if the subject feels less hunger, then the subject should mark X at the second point from far left), taken 180 minutes after having the breakfast with different protein composition
VAS for satiety at 0 minute | baseline
  Visual Analog Scale, a scale in the form of an empty straight line with no values but only several level point (ex: if the line is 10cm, then each cm represent 1 level). Extreme choices are both ends of the straight line. The minimum value is at the left end and the maximum value is at the right end. The subject must make a choice between the two ends of the line by giving an X mark (ex : if the subject feels less hunger, then the subject should mark X at the second point from far left), taken directly after having the breakfast with different protein composition
VAS for satiety at 15 minute | 15 minutes
  Visual Analog Scale, a scale in the form of an empty straight line with no values but only several level point (ex: if the line is 10cm, then each cm represent 1 level). Extreme choices are both ends of the straight line. The minimum value is at the left end and the maximum value is at the right end. The subject must make a choice between the two ends of the line by giving an X mark (ex : if the subject feels less hunger, then the subject should mark X at the second point from far left), taken 15 minutes after having the breakfast with different protein composition
VAS for satiety at 60 minute | 60 minutes
  Visual Analog Scale, a scale in the form of an empty straight line with no values but only several level point (ex: if the line is 10cm, then each cm represent 1 level). Extreme choices are both ends of the straight line. The minimum value is at the left end and the maximum value is at the right end. The subject must make a choice between the two ends of the line by giving an X mark (ex : if the subject feels less hunger, then the subject should mark X at the second point from far left), taken 60 minutes after having the breakfast with different protein composition
VAS for satiety at 120 minute | 120 minutes
  Visual Analog Scale, a scale in the form of an empty straight line with no values but only several level point (ex: if the line is 10cm, then each cm represent 1 level). Extreme choices are both ends of the straight line. The minimum value is at the left end and the maximum value is at the right end. The subject must make a choice between the two ends of the line by giving an X mark (ex : if the subject feels less hunger, then the subject should mark X at the second point from far left), taken 120 minutes after having the breakfast with different protein composition
VAS for satiety at 180 minute | 180 minutes
  Visual Analog Scale, a scale in the form of an empty straight line with no values but only several level point (ex: if the line is 10cm, then each cm represent 1 level). Extreme choices are both ends of the straight line. The minimum value is at the left end and the maximum value is at the right end. The subject must make a choice between the two ends of the line by giving an X mark (ex : if the subject feels less hunger, then the subject should mark X at the second point from far left), taken 180 minutes after having the breakfast with different protein composition

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of Nutrition, Faculty of Medicine Universitas Indonesia, Jakarta, Jakarta Pusat, Indonesia

REFERENCES:
- [Derived] Witjaksono F, Lukito W, Wijaya A, Annisa NG, Jutamulia J, Nurwidya F, Simadibrata M. The effect of breakfast with different macronutrient composition on PYY, ghrelin, and ad libitum intake 4 h after breakfast in Indonesian obese women. BMC Res Notes. 2018 Nov 3;11(1):787. doi: 10.1186/s13104-018-3895-3. PMID 30390699